CLINICAL TRIAL: NCT05468892
Title: Phase II Randomized Study Evaluating the Efficacy of Panitumumab (VEctibix ) and Trifluridine-Tipiracil (LOnsurf) in Pretreated RAS Wild Type Metastatic Colorectal Cancer Patients: the VELO Trial
Acronym: VELO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Fortunato Ciardiello, Principle Investigator, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VELO
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — trifluridine tipiracil drug combination; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Trifluridine-Tipiracil
  Interventions: Drug: Trifluridine Tipiracil
- Arm B (Experimental): Panitumumab + Trifluridine-Tipiracil
  Interventions: Drug: Trifluridine Tipiracil; Drug: Panitumumab 20 MG/1 ML Intravenous Solution [VECTIBIX]

INTERVENTIONS:
Drug: Trifluridine Tipiracil — Trifluridine-Tipiracil will be administered at 35 mg per square meter orally twice daily, with a glass of water within 1 hour after completion of morning and evening meals, 5 days a week, with 2 days of rest, for 2 weeks, followed by a 14-day rest period. One treatment cycle with Trifluridine-Tipiracil consists of the following:
  Days 1-5: Trifluridine / Tipiracil (35 mg/m2/dose) orally twice daily Days 6-7: Rest Days 8-12: Trifluridine / Tipiracil(35mg/m²/dose) orally twice daily Days 13-28: Rest
Drug: Panitumumab 20 MG/1 ML Intravenous Solution [VECTIBIX] — Panitumumab will be administered as a 6 mg/kg intravenous infusion over 60 minutes every 2 weeks (q2w) of a 28-day cycle (Day 1 and Day 15).
  Arms: Arm B

SUMMARY:
This is a randomized phase II, open label, two arm study, evaluating the efficacy of panitumumab in combination with Trifluridine-Tipiracilas third line therapy, after a first line containing an anti-EGFR agent panitumumab(at least 70% of study population) or cetuximab in metastatic colorectal cancer (mCRC) patients.

DETAILED DESCRIPTION:
This is a randomized phase II, open label, two arm study, evaluating the efficacy of panitumumab in combination with Trifluridine-Tipiracilas third line therapy, after a first line containing an anti-EGFR agent panitumumab(at least 70% of study population) or cetuximab. The primary objective is to evaluate the efficacy [as defined by progression free survival (PFS)] of panitumumab in combination with Trifluridine-Tipiracil in pretreated mCRC patients. The secondary objective is to evaluate the objective response rate (ORR), overall survival (OS) and safety. Patients will be randomized in a 1:1 ratio to receive:

Arm A: Trifluridine-Tipiracil Arm B: Panitumumab + Trifluridine-Tipiracil A total of 112 patients will be enrolled. Treatment will be administered in 28-days cycles until disease progression, unacceptable toxicity, withdrawal of consent or death due to any cause.

All patients will be closely monitored for safety and tolerability during all cycles of therapy, at the treatment discontinuation visit, and during the follow-up period. The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 (v. 5.0) will be used to characterize the toxicity profile of the study treatments on all patients. Patients who discontinue treatment for reasons other than disease progression (e.g., toxicity) will continue scheduled tumor assessments until disease progression, withdrawal of consent, study termination by Sponsor, or death, whichever occurs first. In the absence of disease progression, tumor assessments should continue regardless of whether patients start a new anti-cancer therapy, unless consent is withdrawn. All patients will be followed for survival unless consent is withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of colorectal adenocarcinoma
* Diagnosis of metastatic disease
* RAS (NRAS and KRAS exon 2,3 and 4) wild-type in tissue at initial diagnosis
* Efficacy of a first line therapy containing an anti-EGFR agent (panitumumab or ceuximab) with a major response achieved (complete or partial response)
* Progression after a second line therapy
* Available and adequate baseline tumour tissue sample
* Measurable disease according to RECIST criteria v1.1
* Male or female patients > 18 years of age
* ECOG Performance Status 0-1
* Life expectancy of at least 3 months
* Adequate bone marrow, liver and renal function
* If female and of childbearing potential, have a negative result on a pregnancy test performed a maximum of 14 days before initiation of study treatment
* If female and of childbearing potential, or if male, agreement to use adequate contraception (eg, abstinence, intrauterine device, oral contraceptive, or double-barrier method)
* Signed informed consent

Exclusion Criteria:

* Any contraindication to use Trifluridine - Tipiracil or Panitumumab
* More than two previous lines of treatment
* Active uncontrolled infections
* Past or current history of malignancies other than colorectal carcinoma, except for curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix
* Pregnancy
* Breastfeeding
* Interstitial lung disease or pulmonary fibrosis
* Grade III or IV heart failure (NYHA classification)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
PFS | from screening up to 30 months
  PFS: defined as the time from randomization to the earliest documented disease progression or death due to any cause of panitumumab in combination with Trifluridine-Tipiracil vs Trifluridine-Tipiracil"

SECONDARY OUTCOMES:
ORR | from screening up to 30 months
  ORR: per the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 (v1.1), defined as the number of patients achieving an overall best response of complete or partial response divided by the total number of patients
OS | from screening up to 30 months
  OS: defined as the time from randomization to death due to any cause of panitumumab in combination with Trifluridine-Tipiracil vs Trifluridine-Tipiracil
Safety and tolerability analysis: defined as the evaluation of incidence and severity of AEs, graded according to NCI- CTCAE, version 5.0 (v. 5.0). | from screening up to 30 months
  To explore the safety and tolerability of panitumumab in combination with Trifluridine-Tipiracil vs standard third line therapy (Trifluridine-Tipiracil)

CONTACTS AND LOCATIONS:
Overall Officials: Fortunato Ciardiello, Principal Investigator — A.O.U. dell'Università degli studi della Campania "Luigi Vanvitelli"
Locations (8):
- Italy (8):
  - A.O.U. Cagliari - Presidio Policlinico D. Casula, Monserrato, CA
  - A.O.U. Pisana, Pisa, PI
  - A.R.N.A.S. Garibaldi - P.O. GaribaldiNesima, Catania
  - Istituto Europeo di Oncologia, Milan
  - AORN-Ospedale dei colli, UOC Oncologia, Napoli
  - A.O.U. dell'Università degli studi della Campania "Luigi Vanvitelli", Napoli
  - IRCCS Istituto Nazionale Tumori "Fondazione G. Pascale", Napoli
  - Universiyà Campus-Biomedico, Roma

REFERENCES:
- [Derived] Ciardiello D, Martinelli E, Troiani T, Mauri G, Rossini D, Martini G, Napolitano S, Famiglietti V, Del Tufo S, Masi G, Santini D, Avallone A, Pietrantonio F, Lonardi S, Di Maio M, Zampino MG, Fazio N, Bardelli A, Siena S, Cremolini C, Sartore-Bianchi A, Ciardiello F. Anti-EGFR Rechallenge in Patients With Refractory ctDNA RAS/BRAF wt Metastatic Colorectal Cancer: A Nonrandomized Controlled Trial. JAMA Netw Open. 2024 Apr 1;7(4):e245635. doi: 10.1001/jamanetworkopen.2024.5635. PMID 38592721
- [Derived] Napolitano S, Ciardiello D, De Falco V, Martini G, Martinelli E, Della Corte CM, Esposito L, Famiglietti V, Di Liello A, Avallone A, Cardone C, De Stefano A, Montesarchio V, Zampino MG, Fazio N, Di Maio M, Del Tufo S, De Vita F, Altucci L, Marrone F, Ciardiello F, Troiani T. Panitumumab plus trifluridine/tipiracil as anti-EGFR rechallenge therapy in patients with refractory RAS wild-type metastatic colorectal cancer: Overall survival and subgroup analysis of the randomized phase II VELO trial. Int J Cancer. 2023 Oct 15;153(8):1520-1528. doi: 10.1002/ijc.34632. Epub 2023 Jun 30. PMID 37391938
- [Derived] Napolitano S, De Falco V, Martini G, Ciardiello D, Martinelli E, Della Corte CM, Esposito L, Famiglietti V, Di Liello A, Avallone A, Cardone C, De Stefano A, Montesarchio V, Zampino MG, Bordonaro R, Scartozzi M, Santini D, Di Maio M, De Vita F, Altucci L, Marrone F, Ciardiello F, Troiani T. Panitumumab Plus Trifluridine-Tipiracil as Anti-Epidermal Growth Factor Receptor Rechallenge Therapy for Refractory RAS Wild-Type Metastatic Colorectal Cancer: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2023 Jul 1;9(7):966-970. doi: 10.1001/jamaoncol.2023.0655. PMID 37200022